CLINICAL TRIAL: NCT04291300
Title: Lutetium-177-PSMA Radioligand Therapy for Advanced Salivary Gland Cancer, a Phase II Pilot Study.
Brief Title: Lutetium-177-PSMA Radioligand Therapy in Advanced Salivary Gland Cancer Patients
Acronym: LUPSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHN18
Record Dates: First submitted 2020-02-28; First posted 2020-03-02 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Salivary Gland Cancer; Salivary Duct Carcinoma; Adenoid Cystic Carcinoma
MeSH Terms: conditions — Salivary Gland Neoplasms; Carcinoma, Adenoid Cystic

STUDY DESIGN:
Intervention Model Description: Phase II pilot study, single centre, two cohorts. Cohort 1: Patients with R/M ACC Cohort 2: Patients with R/M SDC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lutetium treatment (Experimental): Drug: Lutetium-177-PSMA-I&T, 4 cycles of 7.4 GBq intravenously, every 6 weeks.
  Interventions: Drug: Lutetium-177-PSMA-I&T

INTERVENTIONS:
Drug: Lutetium-177-PSMA-I&T — 4 cycles of 7.4 GBq 177Lu-PSMA every 6 weeks.
  Other Names: Lutetium-177 Prostate Specific Membrane Antigen

SUMMARY:
Phase 2 pilot study, which evaluates the safety and efficacy of Lutetium-177-PSMA radioligand therapy in advanced salivary gland cancer patients.

DETAILED DESCRIPTION:
Rationale: Prostate specific membrane antigen (PSMA) is a transmembrane protein, which is expressed on prostate cancers cells and other malignancies. Recently, several ligands have been developed that target PSMA. Linked to Gallium-68, this enables diagnostic 68Ga-PSMA-PET/CT scans. Linked to Lutetium-177 enables therapeutic 177Lu-PSMA Radioligand therapy. Most research on the diagnostic and therapeutic possibilities of PSMA has been conducted in patients with advanced prostate cancer.

This research group investigates whether these findings also apply to salivary gland cancer (SGC), a rare cancer. Previously the investigators conducted a phase II 68Ga-PSMA imaging study (NCT03319641), to evaluate PSMA ligand uptake in locally advanced, recurrent and metastatic (R/M) ACC and SDC (two subtypes of SGC). A relevant PSMA-ligand uptake was observed in 93% of ACC patients and 40% of SDC patients. Therefore we consider 177Lu-PSMA radioligand therapy a potential new treatment option for these subtypes of SGC.

Objective: To evaluate the safety and efficacy of 177Lu-PSMA RLT in patients with R/M ACC and SDC with PSMA ligand uptake.

Study design: Phase II pilot study, single centre, two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to provide written informed consent.
* Patients must be ≥ 18 years of age.
* Patients must have an ECOG performance status of 0 to 2.
* Patients must have histological, pathological, and/or cytological confirmation of either adenoid cystic carcinoma or salivary duct carcinoma.
* Patients must have incurable, local or regional recurrent or metastatic ACC or SDC.
* Patients with ACC can only participate in case of objective growth in the last three months or complaints due to the disease.
* Patients must have adequate organ function:

  * Sufficient bone marrow capacity as defined by: WBC count (white blood cell) ≥2.5x10^9/L, PLT (platelet) count ≥100x10^9/L, Hb ≥6 mmol/L, absolute neutrophil count (ANC) ≥1.5x10^9/L
  * Adequate liver function as defined by:Total bilirubin ≤1.5 x ULN. For patients known with Gilbert's Syndrome ≤ 3 x ULN is permitted. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 × ULN OR ≤5.0 × ULN for patients with liver metastases.
  * Adequate kidney function as defined by:serum creatinine ≤1.5 x ULN or creatinine clearance ≥ 50 mL/min
* Patients must have measurable disease at baseline. Defined as ≥ 1 lesion ≥ 2 cm (long axis) that is present on baseline CT.
* Patients must have a positive 68Ga-PSMA PET/CT scan, defined by at least one lesion ≥ 1.5 cm (long axis) with a ligand uptake above liver level.

Exclusion Criteria:

* Patients whom are pregnant or breast feeding.
* Patients with reproductive potential not implementing adequate contraceptives measures.
* Patients with known brain metastases or cranial epidural disease or intracardial metastases.
* Patients with concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.
* Patients with urinary tract obstruction or marked hydronephrosis
* Less than 4 weeks since last myelosuppressive therapy or other radionuclide therapy.
* Concomitant cancer treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Adverse events measured using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Through study completion, up until 3 years after last patient commences treatment
  Safety

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, up until 3 years after last patient commences treatment
  Response will be measured according to RECIST version 1.1
Progression free survival (PFS) | Through study completion, up until 3 years after last patient commences treatment
  PFS will be defined as time from study enrollment until disease progression or death.
Overall survival (OS) | Through study completion, up until 3 years after last patient commences treatment
  OS will be defined as time from study enrollment until date of death of any cause.
Duration of response (DoR) | Through study completion, up until 3 years after last patient commences treatment
  Only patients with complete remission or partial response will be included in the assessment of DoR. DoR is defined as time from study enrollment until disease progression or death
Quality of life (QoL) | Trough study completion, up until 3 years after last patient commences treatment
  QoL will be assessed using EORTC QLQ-C30 questionnaire. This is the core questionnaire for assessing health related quality of life of cancer patients participating in clinical trials. It contains 30 items and incorporates a global health status scale, five functional scales, three symptom scales, and several single items assessing additional symptoms. All of the scales and single-item measures range from 0-100. A high score for global health status represents a high QoL, a high score in functional scale represents a high/healthy level of functioning, a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life (QoL) | Trough study completion, up until 3 years after last patient commences treatment
  QoL will be assessed using EORTC QLQ-H&N43 questionnaire. This is an additional questionnaire to assess health related topics relevant for head and neck cancer patients. The module contains 43 questions, all symtom scales or symptom items.All of the scale/item measures range from 0-100. For all scales/items higher scores indicate more problems.
Quality of life (QoL) | Trough study completion, up until 3 years after last patient commences treatment
  QoL will be assessed using performance status scale for head&neck cancer patients (PSS-HN). It contains 3 items, each randing from 0-100. These items are rated by the health professional. A high score indicates a high performance status.
Quality of life (QoL) | Trough study completion, up until 3 years after last patient commences treatment
  QoL will be assessed using pain visual analogue scale (VAS) questionnaire. This include two questions: the average pain during the past week and the worst pain during the past week. Both questions range from 0-100, a higher score indicates more pain.
Dosimetry | From start of study till last patient commences last SPECT/CT (7 days after first treatment cycle)
  Delivered doses will be calculated based on pharmacokinetics in the blood and dosimetry on SPECT/CT imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided